CLINICAL TRIAL: NCT03875846
Title: Intraoperative Simultaneous Pressure Guided Revascularization Study
Acronym: INSTANT
Status: Completed | Type: Observational
Sponsor: Mark Rockley (Other)
Responsible Party: Sponsor-Investigator, Mark Rockley, Study Coordinator, University of Ottawa
Organization: University of Ottawa (Other)
Other Study IDs: 20180656-01H
Record Dates: First submitted 2019-03-13; First posted 2019-03-15 (Actual); Last update posted 2021-08-04 (Actual); Status verified 2021-08

CONDITIONS: Peripheral Vascular Diseases; Blood Pressure; Monitoring, Intraoperative; Clinical Decision-Making; Endovascular Procedures
Keywords: Intraoperative Decision Making; Revascularization; Physiologic Monitoring Feedback
MeSH Terms: conditions — Peripheral Vascular Diseases | interventions — Ankle Brachial Index

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Intraoperative Hemodynamic Improvement: The primary outcome will examine the magnitude of change in the Toe-Brachial Index (TBI) between the beginning and the end of the procedure. The two measurements will be taken before- and after- vascular sheaths had been placed.
  Interventions: Diagnostic Test: Intraoperative Hemodynamic Pressures; Diagnostic Test: Contrast Flow Rate

INTERVENTIONS:
Diagnostic Test: Intraoperative Hemodynamic Pressures — Secondary analyses will examine the Ankle-Brachial Index, and the absolute limb pressures. In addition, the changes in flow rate of contrast before- and after- intervention will be examined as an indicator of perfusion.
  Other Names: Toe Brachial Index; Ankle Brachial Index; Absolute Toe Pressure; Absolute Ankle Pressure
Diagnostic Test: Contrast Flow Rate — A secondary analysis will examine the rate of contrast flow during pre-intervention and post-intervention angiograms, and correlate these findings with hemodynamic measurements recorded during surgery.
  Other Names: Time to Peak Opacification; Rate of Contrast Opacification; Wash-In Rate; Wash-Out Rate

SUMMARY:
This study aims to determine whether intraoperative physiologic measurements of blood flow to the leg during endovascular treatment of Peripheral Arterial Disease (PAD) can predict future clinical outcomes.

DETAILED DESCRIPTION:
Lower extremity peripheral arterial disease (PAD) caused by atherosclerosis can cause cause leg pain, gangrene, and limb loss. PAD is a result of poor blood flow to the extremity, and the emerging most common initial method of interventional treatment is endovascular therapy, for example angioplasty or stenting. The poor blood flow to the extremity can be inferred by the hemodynamic pressure of blood in the leg. These toe or ankle pressure measurements are typically performed before surgery to diagnose PAD, and after surgery as surveillance.

However, endovascular treatment has a high failure rate often exceeding 20% within a year. There is evidence that physiologic measurements prior to treatment and after treatment are closely related to clinical outcomes. This study introduces these physiologic measurements to the operating room, to determine if physiologic improvement can be detected instantaneously during endovascular revascularization. Patients will be followed for a year following surgery to detect hemodynamic and clinical outcomes. The rationale of these intraoperative measurements would be to potentially guide future surgery, by providing real-time hemodynamic feedback to the operator.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing elective or semi-urgent endovascular procedures on lesions of the aorta, iliac, femoral, popliteal, or tibial arteries
* Symptomatic, atherosclerotic Peripheral Vascular Disease. These symptoms include any Rutherford's classification.

Exclusion Criteria:

* Concurrent hybrid open procedure during endovascular revascularization requiring vascular clamping for any period of time, such as endarterectomy
* Prior open vascular surgery performed on the affected leg
* Emergent intervention for Acute Limb Ischemia, defined as symptoms lasting less than 14 days
* Non-femoral vascular access

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing elective or semi-urgent endovascular procedures for lower extremity de-novo atherosclerotic peripheral vascular disease. These patients will be treated at The Ottawa Hospital, Civic Campus, under the care of the Division of Vascular Surgery.
Sampling Method: Non-Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2018-10-01 (Actual); Primary Completion 2020-01-01 (Actual); Study Completion 2021-01-01 (Actual)

PRIMARY OUTCOMES:
Major Adverse Limb Event (MALE) | 1 Year
  Composite outcome of major amputation above the ankle, major re-intervention in the form of catheter-directed thrombolysis, open bypass or thrombectomy.

SECONDARY OUTCOMES:
Major Amputation | 1 Year
  Any ipsilateral leg amputation performed above the joint of the ankle.
Minor Amputation | 1 Year
  Any ipsilateral leg amputation performed distal to the joint of the ankle.
Target Vessel Re-Intervention | 1 Year
  Endovascular, Open, Thrombectomy, Thrombolysis.
Target Vessel Patency | 1 Year
  Primary: Absence of target vessel occlusion or restenosis >50% Primary Assisted: Patency requiring assistance of subsequent procedure to maintain patency of target vessel Secondary: Patency requiring assistance of subsequent procedure to restore patency of target vessel
Improvement in Rutherford's Classification of Peripheral Vascular Disease | 1 Year
  Maximal documented categorical state following index revascularization
Post-Operative Hemodynamic Measurements | 1 - 3 Months
  Correlation between intraoperative completion and immediate post-operative measurements, with longer-term surveillance measurements

OTHER OUTCOMES:
Mortality | 1 Year
  As captured by the hospital's Electronic Health Record
Amputation-Free Survival | 1 Year
  Survival free of major amputation.

CONTACTS AND LOCATIONS:
Overall Officials: George Wells, PhD, MSc, Principal Investigator — Cardiovascular Research Methods Centre, University of Ottawa Heart Institute
Locations (1):
- The Ottawa Hospital, Civic Campus, Ottawa, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Rockley M, Jetty P, Wells GA. Protocol for a prospective observational diagnostic study: intraoperative simultaneous limb pressure monitoring (INSTANT) study. BMJ Open. 2019 Aug 22;9(8):e030456. doi: 10.1136/bmjopen-2019-030456. PMID 31444190